CLINICAL TRIAL: NCT05583045
Title: PREVENT - Prediabetes Intervention With Olive Leaf Tea
Brief Title: Prediabetes Intervention With Tea
Acronym: PREVENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Politécnico de Bragança (Other)
Collaborators: Unidade Local de Saúde do Nordeste (Unknown); European Social Fund (Other)
Responsible Party: Principal Investigator, Manuela Meireles, Principal Investigator, PhD, Instituto Politécnico de Bragança
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 83/2022
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2; Pre Diabetes
Keywords: Olive leaves; Diabetes; Glycaemic control; Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two groups (A or B):
  A: Olive leaf tea + Lifestyle behavior change program B: Placebo tea + Lifestyle behavior change program
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking is from the responsibility of the tea supplier which was asked to send the tea/placebo codified and only reveal the codification after the end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olive Leaf Tea (OLT) (Experimental): Daily intake, for 12 weeks, of olive leaf tea + lifestyle behavior change program.
  Interventions: Other: Olive Leaf Tea; Behavioral: Lifestyle behavior change program (LBC)
- Placebo tea (CON) (Placebo Comparator): Daily intake, for 12 weeks, of placebo tea + lifestyle behavior change program
  Interventions: Behavioral: Lifestyle behavior change program (LBC); Other: Placebo tea

INTERVENTIONS:
Other: Olive Leaf Tea — Olive leaf tea (individual tea bags provided to participants with instructions of preparation)
  Arms: Olive Leaf Tea (OLT)
Behavioral: Lifestyle behavior change program (LBC) — Lifestyle behavior change program as defined by America Diabetes Association on "Standards of Medical Care in Diabetes-2022 Abridged for Primary Care Providers"(Association 2022)
Other: Placebo tea — Placebo tea containing 2,6g cellulose and a caramel coloring
  Arms: Placebo tea (CON)

SUMMARY:
The goal of this interventional study is investigating the effect of the daily consumption of olive leaves tea on glycemic control of individuals diagnosed with pre-diabetes. The hypothesis of this study is that the integration of olive leaf tea on daily food consumption will favors glycemic control and ameliorate insulin resistance in individuals with pre-diabetes.

DETAILED DESCRIPTION:
This study is a triple-blinded, randomized, placebo-controlled trial with parallel assignment

ELIGIBILITY:
Inclusion Criteria:

At least one of three glycemic criteria for pre diabetes as defined by 2022 American Diabetes Association (ADA) guidelines:

* Fasting plasma glucose level, 100 to 125 mg per deciliter (5.6 to 6.9 mml per liter);
* Plasma glucose level 2 hours after a 75-g oral glucose load, 140 to 199 mg per deciliter (7.8 to 11.0 mml per liter);
* Glycated hemoglobin level, 5.7 to 6.4% (39 to 47 mml per mole).

Exclusion Criteria:

* Current use of medication for lowering blood cholesterol, glucose or hypertension;
* History of chronic or severe diseases that may affect study outcomes or limit study participation;
* Pregnancy and breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  Effect of olive leaf tea (OLT) on HbA1c after 12 weeks of intervention in individuals with prediabetes

SECONDARY OUTCOMES:
Fasting Plasma Glicose | 12 weeks
  Effect of olive leaf tea (OLT) on FPG after 12 weeks of intervention in individuals with prediabetes
Insulin | 12 weeks
  Effect of olive leaf tea (OLT) on Insulin after 12 weeks of intervention in individuals with prediabetes
Cholesterol Total, c-HDL, c-LDL and triglycerides | 12 weeks
  Effect of olive leaf tea (OLT) on CT, c-HDL, c-LDL and TG after 12 weeks of intervention in individuals with prediabetes
Aspartate transaminase (AST) and Alanine transaminase (ALT) | 12 weeks
  Effect of olive leaf tea (OLT) on AST and ALT after 12 weeks of intervention in individuals with prediabetes
Alkaline Phosphatase | 12 weeks
  Effect of olive leaf tea (OLT) on Alkaline Phosphatase after 12 weeks of intervention in individuals with prediabetes
Bilirubin | 12 weeks
  Effect of olive leaf tea (OLT) on Bilirubin after 12 weeks of intervention in individuals with prediabetes
Creatinine | 12 weeks
  Effect of olive leaf tea (OLT) on Creatinine after 12 weeks of intervention in individuals with prediabetes

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Meireles, PhD, Principal Investigator — Instituto Politécnico de Bragança
Locations (1):
- Instituto Politécnico de Bragança, Bragança, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All participant data will be collected anonymously and only individual data related to the outcomes will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication of the final results during two years
Access Criteria: Will be available upon request to researcher